CLINICAL TRIAL: NCT04970771
Title: Solving Wellness: An Initiative to Enhance Canadian Healthcare Provider Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Montfort (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-22-06-011
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Stress; Burnout, Professional; Burnout
Keywords: Mental Health; Healthcare Providers; Digital Tools; Wellness Resources
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Solving Wellness Platform Group (Experimental): Participants will receive a 1-year membership to the Solving Wellness virtual platform containing interactive wellness resources.
  Interventions: Behavioral: Solving Wellness platform

INTERVENTIONS:
Behavioral: Solving Wellness platform — Interactive wellness resources available include a wide range of curated content and resources including fitness and yoga classes, cooking classes, webinars on sleep and various mental health topics including resilience, stress management, relationships and mindfulness, and resources including e-books, videos and guided meditations. Online discussion groups will foster awareness for specific issues and allow casual discussion. A curated collection of links to additional resources including the Solving Healthcare podcast will also be provided.

SUMMARY:
Given the high incidence of burnout, depression, and suicidal ideation among Canadian healthcare providers (HCPs), there is an urgent need to support wellness through strengthening peer networks and engaging key stakeholders. This project will explore the capacity of digital tools to educate HCPs and enable them to support their mental health. The investigators will evaluate specific research questions: Are HCPs more aware of their wellness needs? Did burnout and stress decrease? Do HCPs feel more supported by their peers? The overarching objective is to contribute towards a culture prioritizing HCP wellbeing. The investigators hope to achieve this through two outcome-oriented objectives: 1) to create resources to promote HCP wellbeing and 2) to foster a web-based HCP community. This initiative integrates big data tools, interactive online content, and the Solving Healthcare podcast to improve HCP wellness. It is anticipated that HCPs will become more aware of their wellness needs, and once they are able to identify strategies to live healthier work lives, cultural changes will take place, leading to a new attitude surrounding HCP mental health. To complete these objectives, resources will be drawn from the HELP-MD physician database and an advisory circle, and will be disseminated via a web platform and the widely known Solving Healthcare podcast. The project's significance stems from the changes it will incite in both individuals and health care institutions, inspiring long term changes in workplace culture and teaching the next generation that a balanced work life is attainable.

ELIGIBILITY:
Participant Inclusion Criteria Healthcare providers who are

* aged 18 years or older
* physicians, residents, medical students, nurses, and allied health professionals of various specialties at the Montfort Hospital and will also be open to Canadian medical professionals (physicians, residents, medical students, nurses, and allied health professionals).

Participant exclusion criteria: Healthcare providers who have previously enrolled as a member of Solving Wellness prior to project start.

Stakeholder staff inclusion criteria:

Employees who are

* aged 18 years or older; and
* whose roles provide them with direct knowledge of topics relating to physician wellness at the Montfort Hospital and of the interventions implemented during the study period (e.g., senior physicians, experts on physician wellness, health system decision makers, mental health experts, health care service managers, nurse managers, ICU managers, medical site lead, directors or department heads).

Stakeholder staff exclusion criteria: Any employees who are involved in the project design and execution (ie. advisory circle members or research team members)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in healthcare provider burnout | 12 months
  As measured by the administration of the Maslach Burnout Inventory (MBI) at Months 1 and 12 of the intervention phase. The MBI is a 22 question survey which evaluates 3 subscales; emotional exhaustion, depersonalization and reduced personal accomplishment. Each question is rated from 1 to 5, where 1 is strongly disagree and 5 is strongly agree. A high score on the emotional exhaustion subscale (27+) coupled with a high score on the depersonalization scale (10+) indicates that the individual may be experiencing 1+ symptoms of burnout.
Reduction in healthcare provider stress | 12 months
  As measured by the administration of the Perceived Stress Scale (PSS) at Months 1 and 12 of the intervention phase. The PSS consists of 10 questions, answered on a scale of 0-4 depending on the frequency of which the behavior is observed, with 0 indicating "never" and 4 indicating "very often". Overall, a score of 0 indicates low stress, while a score of 40 indicates an individual with high perceived stress levels.
Increase in perceived peer support | 12 months
  A pre/post intervention staff questionnaire will measure this outcome quantitatively through the inclusion of questions relating to the degree of perceived peer support , and measured qualitatively by thematic analysis of post-intervention focus group discussions with study participants and staff stakeholders.
Increased awareness of personal wellness needs | 12 months
  A pre/post intervention staff questionnaire will measure this outcome quantitatively through the inclusion of questions relating to the degree that wellness is considered daily, and measured qualitatively by thematic analysis of post-intervention focus group discussions with study participants and staff stakeholders.
Increased ability to apply wellness practices to daily life | 12 months
  A pre/post intervention staff questionnaire will measure this outcome quantitatively through the inclusion of questions relating to the degree that wellness is considered daily, and qualitatively measured by thematic analysis of post-intervention focus group discussions with study participants and staff stakeholders.

CONTACTS AND LOCATIONS:
Overall Officials: Kwadwo Kyeremanteng, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- Montfort Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No